CLINICAL TRIAL: NCT03951818
Title: Observing the Changes of Endocrine and Metabolism in Patients With Thalassemia Major
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201903041RINB
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patient with thalassemia major have many endocrine diseases, such as hypopituitarism, hypothyroidism, hypoparathyroidis, osteoporosis, and etc.. These problems may be due to anemia itself or related to iron deposition. This study aimed to investigate the endocrine aspect of thalassemia major patients in Taiwan in order to introduce early intervention or treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Thalassemia major
* Patients of 20-85 years old

Exclusion Criteria:

* Patients younger than 20 years old.
* Patients older than 85 years old.
* Patients who are pregnant

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20-85 years old thalassemia major patients treated in the OPD of NTUH
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Abnormal bone mineral density rate | 10 years
  abnormal bone mineral density is defined as T-score < -1 SD in menopause women or men older than 50 years old, or Z score < -2 SD in premenopausal women or men not older than 50 year old.

SECONDARY OUTCOMES:
abnormal thyroid function rate | 10 years
  abnormal thyroid function is defined as abnormal free thyroxine or abnormal thyrotropin. Normal range of free thyroxine is 0.6-1.75 ng/dl. normal range of thyrotropin is 0.1-4.5 mU/l.
abnormal pituitary function rate | 10 years
  abnormal pituitary function is defined as any of the abnormality in serum adrenocorticotropin (pg/l), IGF-1 (ng/ml). thyrotropin (mU/l), FSH (U/l), LH (U/l)

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Shyang-Rong Shih, Taipei, Taiwan

REFERENCES:
- [Derived] Yang WP, Chang HH, Li HY, Lai YC, Huang TY, Tsai KS, Lin KH, Lin DT, Jou ST, Lu MY, Yang YL, Chou SW, Shih SR. Iron Overload Associated Endocrine Dysfunction Leading to Lower Bone Mineral Density in Thalassemia Major. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz309. doi: 10.1210/clinem/dgz309. PMID 31907538